CLINICAL TRIAL: NCT06452394
Title: NEODOXy: Targeting Cancer Stem Cells With NEOadjuvant DOXYcycline in Patients With Early Estrogen Receptor Positive / Human Epidermal Growth Factor Receptor 2- Negative Breast Cancer. A Prospective, Multicenter, Single Arm, Open Label Phase II Trial
Brief Title: NEODOXy: Targeting Breast Cancer Stem Cells With Doxycycline
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 21/23
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: early ER+/HER2- breast cancer; NEODOXy; Doxycycline; Human Epidermal Growth Factor Receptor 2 negative; Estrogen Receptor; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: A prospective, single arm, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEOadjuvant DOXYcycline (Experimental): neoadjuvant chemotherapy (4 cycles epirubicin 90 mg/m2 + cyclophosphamide 600 mg/m2 q3W followed by 4 cycles weekly paclitaxel (D1, D8, D15) 80 mg/m2)
  + doxycycline (200 mg/day from D5 to D18 of each cycle)
  Interventions: Drug: Doxycyclin

INTERVENTIONS:
Drug: Doxycyclin — Belongs to the class of tetracyclines. It has bacteriostatic activity against a broad range of gram-positive and gram-negative bacteria. Its mechanism of action lies in the binding to the 30S ribosomal subunit
  Other Names: Doxyclin

SUMMARY:
Despite modern surgical and medical treatments, breast cancer can re-occur and lead 20% of patients to death. During the last 20 years, pre-clinical studies have shown that treatment failures may be due to the presence of a sub-type of cancer cells, the cancer stem cells, which are resistant to chemotherapy and radiotherapy. By chance, doxycycline, an old, inexpensive and safe molecule seems to target effectively these cancer stem cells. This study proposes to check for the clinical efficacy of doxycycline to target the cancer stem cells and improve the response to neoadjuvant chemotherapy in ER+/HER2- breast cancers.

DETAILED DESCRIPTION:
Patients with early stage ER+/HER2- breast cancer (BC) have a low pathologic complete response (pCR) rate of less than 15%. Over the past 20 years, studies have identified a subset of cancer cells with tumorigenic and stem-like properties, known as cancer stem cells (CSCs), that are involved in tumour initiation, metastasis, relapse and resistance to treatment. Cancer cells with stem-like properties are known to possess cellular plasticity that not only enables self-renewal capacity, but also exhibits high tumourigenic potential and resistance to oncological therapies such as chemotherapy and/or radiotherapy.

CSCs can arise from normal adult breast stem cells through mutations or directly from differentiated tumor cells. Tumour hypoxia has been shown to be one of the major factors promoting and maintaining the stemness phenotype. The metabolism of CSCs in hypoxia relies on a delicate balance between reduced energy requirements through reduced proliferation and an altered balance between mitochondrial oxidative phosphorylation ("OXPHOS") and cytosolic glycolysis, while maintaining mitochondrial redox homeostasis to control reactive oxygen species (ROS) levels. Any slight imbalance in mitochondrial redox homeostasis in CSCs, leading to transient effects on ROS, may promote their differentiation towards their non-stem tumour cell counterparts. Consequently, specific drugs targeting mitochondrial metabolism, leading to increased ROS levels, may destabilise CSCs.

This study proposes to check for the clinical efficacy of doxycycline to target the cancer stem cells and improve the response to neoadjuvant chemotherapy in ER+/HER2- breast cancers. The change in the stemness marker, ALDH1, assessed before and after treatment and the effect of doxycycline on the pathological response will be studied.

The translational work will be to better define these stem cells and to grow organoid cultures to study the effects of the different drugs in vitro. This study also aims to address a number of translational research questions using a tumor sample obtained from an additional core biopsy prior to treatment initiation and using a fresh tumor sample from the surgical specimen in the case of residual tumor after neoadjuvant treatment:

* Quantify and characterise the effects of doxycycline on tumors
* Identify factors that facilitate or prevent the effects of doxycycline
* Estimate the effect of doxycycline compared to other CSC-targeting drugs

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and current ICH GCP E6 regulations before registration and prior to any trial specific procedures.
* Histologically confirmed ER+/HER2- primary invasive breast cancer, according to ASCO/CAP Guideline1,2, defined as ER expression rate ≥ 1%.
* Patients are candidate for curative surgery and with a tumor size of at least 2 cm and nodal classification cN0-3 according to the 8th edition, January 2017 of the anatomic TNM classification3.
* Patients with multiple synchronous ipsilateral tumors are allowed, as long as all lesions are ER+/HER2-. Only one target lesion will be considered for ALDH1 primary endpoint, and the target lesion has to be the largest lesion.
* Patients are planned for neoadjuvant chemotherapy according to the local standards.
* Patients accept standard curative surgery after neoadjuvant chemotherapy with 4 cycles of epirubicin and cyclophosphamide (EC) followed by 12 doses of weekly paclitaxel (or nab-paclitaxel).
* Diagnostic tumor tissue is available for the mandatory central pathology examinations; or an additional biopsy is planned in case of lack of remaining material from the diagnostic biopsy, provided that the patient has consented to the optional TR-project.
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration in this trial and the patient has no evidence of disease at registration. Less than 2 years is acceptable for adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Male or female patients age ≥ 18 years.
* ECOG performance status 0-1.
* Adequate bone marrow function:

  * neutrophil count ≥ 1.5 x 10^9/L,
  * platelet count ≥ 100 x 10^9/L,
  * hemoglobin ≥ 90 g/L.
* Adequate hepatic function:

  * total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease max. 3.0 x ULN),
  * AST and ALT ≤ 2.5 x ULN.
* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73 m2 (according to CKD-EPI formula).
* No known cardiac dysfunction contraindicating the planned neoadjuvant chemotherapy with 4 cycles of EC followed by 12 doses of weekly paclitaxel.
* Women of childbearing potential must use highly effective, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 12 months after the last dose of investigational drug. A negative pregnancy test before inclusion into the trial is required for all women of childbearing potential.
* Men agree not to donate sperm or to father a child during trial treatment and until 12 months after the last dose of investigational drug.
* Patient is able and willing to swallow trial drug as whole tablet.

Exclusion Criteria:

* Patients with 2 synchronous breast cancers or more of different subtypes (other than ER+/HER2-).
* Metastatic patients.
* Patients having received or planned to undergo neoadjuvant endocrine therapy or other investigational therapies before surgery.
* History of intracranial hypertension (IH).
* Concomitant or recent (within 30 days of registration) treatment with any other experimental drug.
* Concomitant use of drugs contraindicated with doxycycline according to the Swissmedic-approved product information or contraindicated according to the trial protocol.
* Use of dietary supplements, natural therapies, phytotherapy or complementary and integrative medicines (homeopathy, spagyric remedies, etc) without approval of the sponsor.
* Concomitant use of other anti-cancer drugs or radiotherapy.
* Patients having received doxycycline or other antibiotics of the cyclin family within 28 days before registration.
* Known hypersensitivity to cyclin group of substances, including tetracyclines, doxycycline or to any component of the trial drug.
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the proportion of patients with ALDH1 positive tumors before and after neoadjuvant chemotherapy plus doxycycline. | From the date of registration to 30 days after last trial treatment
  Difference in the proportion of patients with Aldehyde Dehydrogenase 1 (ALDH1) positive tumors before and after neoadjuvant chemotherapy plus doxycycline, assessed as follows: Tumor cells expressing ALDH1 will be revealed by immunostaining using an anti-ALDH1 antibody on the pathology slides. In case of residual disease, an ALDH1 positive tumor is defined as having at least 5% of its tumor cells expressing ALDH1. In case of pCR, determined by H&E staining, ALDH1 will be considered negative.
Pathologic complete response rate after surgery, defined as no invasive residual disease in the breast and in the axillary lymph nodes. | From the date of registration to 30 days after last trial treatment
  Pathologic complete response (pCR) rate after surgery in the breast and in the axillary lymph nodes (if biopsy-proven lymph node involvement prior to neoadjuvant treatment), defined as proportion of patients with no residual invasive cancer for each anatomic location (i.e no viable cancer cell on microscopic examination after Hematoxylin and Eosin (H&E) staining): ypT0-ypTis ypN0.

SECONDARY OUTCOMES:
Percentage of ALDH1 positive tumor cells | From the date of registration to 30 days after last trial treatment
  Difference in the percentage of ALDH1 positive tumor cells before and after neoadjuvant chemotherapy plus doxycycline
Difference in the percentage of ALDH1 positive tumor cells | From the date of registration to 30 days after last trial treatment
  Category of the difference in the percentage of ALDH1 positive tumor cells before and after neoadjuvant chemotherapy plus doxycycline
Pathological residual disease | From the date of registration to 30 days after last trial treatment
  Pathological residual disease using the validated residual cancer burden score (RCB score)
Radiological tumor shrinkage | From the date of registration to 30 days after last trial treatment
  Radiological tumor shrinkage at mid-term and at completion of neoadjuvant treatment
Breast conservation rate | From the date of registration to 30 days after last trial treatment
  Breast conservation rate at surgery and the rate of conversion from mastectomy to breast conserving surgery
Doxycycline adherence rate | From the date of registration to 30 days after last trial treatment
  Doxycycline adherence rate
Patient-reported treatment burden | From the date of registration to 30 days after last trial treatment
  Patient-reported treatment burden and satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Lelièvre, M.D., Study Chair — Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (8):
- Switzerland (8):
  - Kantonsspital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Clinique de Genolier, Genolier, Canton of Vaud
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Tumor Zentrum Aarau, Aarau
  - Réseau du sein Lausanne, Lausanne
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Tumor- und Brustzentrum Ostschweiz, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No
The translational work will be to better define these stem cells and to grow organoid cultures to study the effects of the different drugs in vitro and will be carried out as part of this trial. Only data from patients who agreed to an additional biopsy of tumour tissue will be used for translational research.